CLINICAL TRIAL: NCT03460054
Title: The SPOR Canadian Glomerulonephritis Registry and Translational Research Initiative
Brief Title: The Canadian Glomerulonephritis Registry and Translational Research Initiative
Acronym: CGNR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Providence Health & Services (Other); Foothills Medical Centre (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Queen Elizabeth II Health Sciences Centre (Other); CHU de Quebec-Universite Laval (Other); The Ottawa Hospital (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: CAPCR 16-6110
Record Dates: First submitted 2018-02-16; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Glomerular Nephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — DNA, serum, plasma, urine and throat swabs will be obtained from patient at each research visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- IgA Nephropathy (IgAN): Biopsy-Proven IgAN
- Focal Segmental Glomerulosclerosis (FSGS): Biopsy-Proven FSGS
- Membranous Nephropathy (MGN): Biopsy-Proven MGN
- Mesangioproliferative Glomerulonephritis (MPGN): Biopsy-Proven MPGN
- Minimal Change Disease (MCD): Biopsy-Proven MCD

SUMMARY:
Glomerulonephritis (GN) is one of the most important causes of kidney failure in Canada. These comprise a group of "rare" diseases (<5 per 250,000 population), yet GN is a leading cause of kidney failure and accounts annually for close to 20% of incident cases of end stage kidney disease (ESKD) in Canada. Prevention of progression to kidney failure is possible, however several barriers and gaps in knowledge challenge our ability to provide patients with individualized effective therapy. These include a lack of sensitive non-invasive tools for monitoring disease activity, prognosis, and response to therapy. A gap in understanding of the core molecular processes underlying the development and progression of GN, and a lack of cohesive networks for evaluation of novel treatment approaches contribute to a lack of targeted and personalized therapies for GN. To address these challenges we will create a national, multi-dimensional platform for application of human-based molecular research and advanced therapeutics in GN.

DETAILED DESCRIPTION:
To accomplish the goals set out in this project, the CGNR network will recruit and maintain a large cohort of patients 350 with glomerular diseases and follow them prospectively with standardized clinical data and biospecimen collection. The infrastructure and study design presented in this protocol will form the backbone for a broad range of scientific approaches and inquiries, essential to moving the field forward and improving the outcomes of patients affected by these diseases. Successful recruitment of 350 patients from across the country, creating a rich biobank and data repository. Our aims are to identifying patient characteristics associated with glomerular diseases and complications, characterizing disease trajectory under current clinical care, estimating event rates of clinically meaningful outcomes, identify predictors of short and long-term outcomes including therapeutic outcomes. We also aim to identify and characterize clinical, histological, molecular and genetic biomarkers that are linked to glomerular diseases and outcomes that might improve disease classification, and biomarkers that may be employed in clinical practice or in clinical trials that predict disease activity or response to therapy. Furthermore, we propose to study sequence variations, transcriptome profile and their impact on disease presentation and clinical outcome. On the patient level, we will identify patient reported outcomes such as disease burden, physical function and quality of life associated with GN diseases and validate tools to assess impact of disease and therapy on patients. Achievement of our goals will be determined by the success of the research studies that evolve from the biobank, and data repository.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IgAN, FSGS, MCD, MGN, MPGN
* age 18-80 inclusive
* estimated GFR>=30ml/min/1.73m2 estimated using 4 variable MDRD
* first kidney biopsy within 12 months of enrollment
* connective tissue disease serology is normal/negative ANA, ANCA

Exclusion Criteria:

* Systemic lupus erythematosus (SLE) - serology supported
* Evidence of diabetic nephropathy on renal biopsy
* Underlying connective tissue disease and/or serologic evidence (sarcoid, rheumatoid arthritis, vasculitis)
* Prior organ transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patient who has biopsy proven IgAN or FSGS, MCD, MGN, MPGN with kidney function GFR>=30
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite renal outcome (Estimated Glomerular Filtration Rate) | 2 years
  End Stage Renal Disease (eGFR<15 or dialysis>60 days) or 40% decline in GFR at 2 years

SECONDARY OUTCOMES:
Rate of renal function decline | 2 years
  slope of least-squares regression line calculated for each person over 2 years
Complete remission of proteinuria | 2 years
  proteinuria <0.3g/day
Partial remission of proteinuria | 2 years
  Defined by % reduction in 24 hour protein excretion from peak value

CONTACTS AND LOCATIONS:
Overall Officials: Heather Reich, MD, Principal Investigator — Nephrologist
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hildebrand AM, Barua M, Barbour SJ, Tennankore KK, Cattran DC, Takano T, Lam P, De Serres SA, Samanta R, Hladunewich MA, Fairhead T, Poyah P, Bush DD, MacLaren B, Sparkes D, Boll P, Jauhal A, John R, Avila-Casado C, Reich HN. The Canadian Glomerulonephritis Registry (CGNR) and Translational Research Initiative: Rationale and Clinical Research Protocol. Can J Kidney Health Dis. 2022 Apr 8;9:20543581221089094. doi: 10.1177/20543581221089094. eCollection 2022. PMID 35450151